CLINICAL TRIAL: NCT02924792
Title: Sternal Intraosseous Transfusion of Autologous Whole Blood: A Comparison of Flow Rates and Degree of Hemolysis
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Ministry of Defence, Norway (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2014/691
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-10

CONDITIONS: Hypovolemic Shock; Hemorrhagic Shock
Keywords: Intraosseous access
MeSH Terms: conditions — Shock; Shock, Hemorrhagic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Reinfusion - Fast1: Case: Autologous reinfusion through Fast1 sternal needle. (Pyng Medical) CE marked/FDA Approved
  Interventions: Device: Reinfusion - Sternal IO needle
- Reinfusion - T.A.L.O.N: Case: Autologous reinfusion through T.A.L.O.N sternal needle. (Vidacare) CE Marked/FDA approved
  Interventions: Device: Reinfusion - Sternal IO needle
- Reinfusion - Intravenous line: Control: Autologous reinfusion through standard intravenous line
  Interventions: Device: Reinfusion - Intravenous needle

INTERVENTIONS:
Device: Reinfusion - Sternal IO needle
  Groups: Reinfusion - Fast1; Reinfusion - T.A.L.O.N
Device: Reinfusion - Intravenous needle
  Groups: Reinfusion - Intravenous line

SUMMARY:
In this study the impact of two CE marked and FDA approved sternal needles in comparison to intravenous access on the flow-rate of autologous reinfusion of whole blood and the possible hemolysis of red cells post-transfusion in a population of healthy military officers is investigated.

DETAILED DESCRIPTION:
Intraosseous (IO) access is an old technique for achieving entrance to the systemic circulation, which has gained resurgence in the last 30 years.

Whether due to trauma or disease, vascular collapse may delay or preclude even experienced medical providers from obtaining standard intravenous (IV) access. Access to the vascular system of the critically ill or injured adult or pediatric patient is essential for resuscitation, and flow rates close up to what can be obtained by using intravenous access is preferable in patient needing immediate fluid boluses for shock resuscitation. Intraosseous access takes advantage of the vascularity of cancellous bone, the spongy bone inside the hard, and access to the highly vascular intramedullary space of bones provides a direct link to central circulation. In addition to using long bones, the sternum is used for intraosseous access and has gained increased use especially in combat casualty care.

However, in a recent publication, the intraosseous route used for transfusion of blood components is questioned. Based on theoretical models for flow rates through porous media and personal clinical observations the authors conclude that the maximum flow rates attainable for transfusion of blood via intraosseous route are inadequate for successful resuscitation. They also fear that additional pressure needed to obtain adequate flow rate may cause hemolysis of red blood cells. Further they postulate that as the bone mineral density reaches a peak occurring in the early 20s, and that a small increase in bone density may cause exponential decrease in intrinsic permeability, there could be a 10-fold decrease in permeability in military age causalities compared to the elderly. The critical points highlighted in this review are in great contrast to recent experience with the use of sternal and humeral I.O's in Operation Enduring Freedom (OEF).

This observational study investigates the impact of two CE marked and FDA approved sternal needles in comparison to intravenous access on the flow-rate of autologous reinfusion of whole blood and the possible hemolysis of red cells post-transfusion in a population of healthy military officers. We also investigate the technical success rate of sternal IO Access between two CE marked and FDA approved sternal Devices. As a supplementary investigation we seek to investigate the anatomic changes as shown by Magnetic Resonance Imaging in individuals who have received multiple intraosseous sternal needles With autologous reinfusion of whole blood.

ELIGIBILITY:
Inclusion Criteria:

* Male, Professional special forces military officers
* Medically cleared for for military exercise or Activity
* Signed standardized informed consent

Exclusion Criteria:

* Participants who will not provide informed consent

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy military officers
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Flowrate of reinfusion of whole blood | 45 minutes
  The total time of reinfusion of 450cc Whole blood
Post transfusion hemolysis | 3 hours
  Hemolysis as measured by Haptoglobin and LD measures

SECONDARY OUTCOMES:
Success rate of sternal IO access | 30 minutes
  The success rate of a valid IO Access, evaluated by expret

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available within 6 months of study completion.